CLINICAL TRIAL: NCT02843165
Title: Randomized Phase II Study of Checkpoint Blockade Immunotherapy Combined With Stereotactic Body Radiation Therapy in Advanced Metastatic Disease
Brief Title: Checkpoint Blockade Immunotherapy Combined With Stereotactic Body Radiation in Advanced Metastatic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Andrew Sharabi, Assistant Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151570
Record Dates: First submitted 2016-07-14; First posted 2016-07-25 (Estimated); Results first posted 2025-07-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Cancer
Keywords: stereotactic body radiation therapy; checkpoint blockade immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Checkpoint blockade immunotherapy plus SBRT (Experimental): Checkpoint blockade immunotherapy (CBI) plus stereotactic body radiation therapy (SBRT)
  Interventions: Radiation: Checkpoint blockade immunotherapy plus SBRT
- Checkpoint blockade immunotherapy (Active Comparator): Checkpoint blockade immunotherapy (CBI) alone
  Interventions: Drug: Checkpoint blockade immunotherapy

INTERVENTIONS:
Drug: Checkpoint blockade immunotherapy — Approved Checkpoint blockade immunotherapy (including anti-CTLA-4 and anti-PD-1/PD-L1 antibodies)
  Arms: Checkpoint blockade immunotherapy
Radiation: Checkpoint blockade immunotherapy plus SBRT — SBRT at 28.5 Gy (9.5 Gy x3 fractions) will be delivered within 1 - 21 days of the start of Cycle 1 of the CBI plus CBI (approved CBIs including anti-CTLA-4 and anti-PD-1/PD-L1 antibodies)
  Arms: Checkpoint blockade immunotherapy plus SBRT

SUMMARY:
The purpose of this study is to determine whether stereotactic body radiation therapy (SBRT) combined with checkpoint blockaded immunotherapy (CBI) will improve the response to the anticancer treatment compared to CBI alone in patients with advanced metastatic cancer.

DETAILED DESCRIPTION:
Patients who will receive anti-PD-1/PD-L1 immunotherapy with at least 1 site of measurable metastatic disease which will not be irradiated will be candidates for the study. Patients will be randomized (1:1) to CBI combined with SBRT or CBI alone. SBRT at 9.5Gy x3 fractions will be delivered within 1-21 days of the start of first cycle of CBI. The first six patients will be treated and observed for toxicity in the safety run-in phase for 30 days after radiation before continuing with further accrual. Radiation dose reduction is allowed if necessary to meet tissue constraints (6Gyx3 Minimum Dose). Response rates will be determined from the non-irradiated lesion/lesions. Blood draws will be obtained to analyze anti-tumor immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Patient has one lesion that is treatable with SBRT.
* Patient has at least 1 site of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria on computed tomography (CT) or Magnetic resonance imaging (MRI) which will not be irradiated.
* Histological confirmation of malignancy (primary or metastatic tumor).
* Patient may have any prior therapy allowed aside from having had prior radiotherapy to the treatment site.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient's screening laboratory values must meet protocol limits.
* Patient must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patient has had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patient receiving any investigational or experimental agents other than immunotherapy.
* Patient who has had any prior radiotherapy to the treatment site(s).
* Patient is a pregnant woman (pregnant women are excluded from this study because radiation treatment has known potential for teratogenic or abortifacient effects).
* Patient refuses to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sharabi, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Moores Cancer Center of the University of California San Diego
Period: Overall Study
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
Started | 58 | 48
Completed | 58 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy | Total
Number analyzed (Participants) | 58 | 48 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.03 (12.9) | 63 (13.5) | 61.92 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 28 | 25 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 49 | 39 | 88
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 4 | 7
  White | 38 | 30 | 68
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 48 | 106
Body System [Count of Participants; unit: Participants] — Cancer type (body system)
  Participants
    Breast | 2 | 3 | 5
    Gastrointestinal | 22 | 24 | 46
    Genitourinary | 6 | 5 | 11
    Gynecologic | 11 | 9 | 20
    Head and Neck | 12 | 1 | 13
    Musculoskeletal | 1 | 2 | 3
    Respiratory | 1 | 2 | 3
    Skin | 1 | 1 | 2
    Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Responses measured by RECIST at 16 weeks from baseline
Population: All participants who received at least one cycle of checkpoint blockade immunotherapy with or without SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
Number analyzed (Participants) | 58 | 48
Participants | 11 | 6

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events assessed from time of first dose to treatment completion (approximately 1 year)
Time Frame: up to 5 years
Population: All participants who received at least one cycle of checkpoint blockade immunotherapy with or without SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
Number analyzed (Participants) | 58 | 48
Participants | 58 | 48

3. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Assessed at 5 years
Population: All participants who received at least one cycle of checkpoint blockade immunotherapy with or without SBRT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
Number analyzed (Participants) | 58 | 48
months | 2.38 [1.95 to 3.37] | 1.88 [1.82 to 2.81]

4. Secondary Outcome: Overall Survival
Description: The time from starting treatment until death due to any cause.
Time Frame: Assessed at 5 years
Population: All participants who received at least one cycle of checkpoint blockade immunotherapy with or without SBRT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
Number analyzed (Participants) | 58 | 48
months | 14.1 [8.46 to 25.2] | 12.6 [7.14 to 29.2]

5. Secondary Outcome: Rate of Stable Disease
Description: The rates of stable disease great than or equal to 6 months during and after SBRT in combination with CBI compared to CBI alone.
Time Frame: Assessed at 5 years
Population: All participants who received at least one cycle of checkpoint blockade immunotherapy with or without SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
Number analyzed (Participants) | 58 | 48
Participants | 7 | 4

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Checkpoint Blockade Immunotherapy Plus SBRT | Checkpoint Blockade Immunotherapy
All-Cause Mortality (participants affected / at risk) | 36/58 | 29/48
Serious Adverse Events (participants affected / at risk) | 24/58 | 15/48
Other Adverse Events (participants affected / at risk) | 44/58 | 35/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Checkpoint Blockade Immunotherapy Plus SBRT (N=58) | Checkpoint Blockade Immunotherapy (N=48)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (4)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Edema limbs (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 2 (2)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Checkpoint Blockade Immunotherapy Plus SBRT (N=58) | Checkpoint Blockade Immunotherapy (N=48)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (4) | 1 (2)
CARDIAC DISORDERS (Cardiac disorders) | 5 (8) | 2 (2)
EAR AND LABYRINTH DISORDERS (Ear and labyrinth disorders) | 3 (4) | 2 (2)
ENDOCRINE DISORDERS (Endocrine disorders) | 6 (6) | 4 (5)
EYE DISORDERS (Eye disorders) | 3 (3) | 2 (2)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 23 (45) | 15 (19)
GENERAL DISORDERS (General disorders) | 21 (33) | 16 (30)
IMMUNE SYSTEM DISORDERS (Immune system disorders) | 1 (1) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 3 (4) | 7 (7)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INVESTIGATIONS (Investigations) | 9 (20) | 6 (14)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 8 (12) | 3 (4)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS (Musculoskeletal and connective tissue disorders) | 15 (23) | 6 (9)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 8 (9) | 3 (4)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 5 (5) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 4 (4) | 2 (2)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 1 (1) | 2 (3)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 12 (22) | 7 (9)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 16 (26) | 13 (14)
VASCULAR DISORDERS (Vascular disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT02843165/Prot_SAP_000.pdf